CLINICAL TRIAL: NCT07179198
Title: A Prospective, Multicenter, Randomized, No-Treatment-Controlled, Assessor-Blinded, Superiority Clinical Investigation to Evaluate the Safety and Effectiveness of Kytogen Defend in Facial Skin Quality Improvement
Brief Title: A Study to Evaluate the Safety and Effectiveness of Kytogen Defend in Facial Skin Quality Improvement in Adult Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinclair Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XKL-CT001-CIP
Record Dates: First submitted 2025-09-03; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Skin Quality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KIO021 - Arm 1 (Experimental)
  Interventions: Device: KIO021
- N/A - Arm 2 (No Intervention)

INTERVENTIONS:
Device: KIO021 — KIO021 is used as a device product for dry skin and dull complexion
  Arms: KIO021 - Arm 1

SUMMARY:
This study was designed to evaluate the efficacy and safety of KIO021, an injectable solution for carboxymethyl chitosan, for temporary improvement of facial skin condition. Designed for forward-looking effectiveness.

To achieve this, it is planned that 500 subjects with dry skin and dull complexion on the face will be included in the injection.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects ≥18 years (subject to the time of signing the ICF), without any restriction on gender; (2) Skin types ranging from type II to IV according to Fitzpatrick classification; (3) The subject exhibits symptoms of dry skin and dull complexion on face, and has a temporary need to improve the quality of facial skin. After evaluation by the investigator, it is deemed suitable for improvement through the medical device used in this trial;

Exclusion Criteria:

* (1) Subjects who have known allergies to Carboxymethyl Chitosan Solutions or any ingredients contained in the product; have known allergies to any local anesthetics (e.g., lidocaine or other amide-type anesthetics) or to an excipient of 5% EMLA cream; are allergic to chlorhexidine (or similar products) or to an excipient found in 0.5% alcohol chlorhexidine; or have a history of severe allergies or any episodes of anaphylactic shock; (2) Subjects having participated in other clinical trials within 1 month prior to enrollment in this trial or being currently participating in other clinical trials; (3) Females who are pregnant, breastfeeding, or planning to become pregnant during the study, or those who have been menopausal for less than 1 year or are in the perimenopausal phase without undergoing hormone therapy; (4) Subjects who have been exposed to strong sunlight or strong ultraviolet rays within 1 month before screening, or who are expected to work outdoors for a long time or need to be exposed to strong sunlight or ultraviolet rays during the study period; (5) Having tattoos, piercings, significant facial hair, scars, deformities, unhealed wounds, active skin diseases or inflammation or infections (e.g., herpes, acne, eczema, dermatitis, psoriasis, herpes zoster, mycosis and papillomas, etc.), abscess, granuloma, active or persistent perinasal infection, cancers or precancerous lesions, malignant tumours or skin swellings with unknown nature, unknown injections, and facial subcutaneous fixations (mesh, thread, gold twisted wire), etc. in the injection and evaluation area that may affect the effectiveness evaluation or increase treatment-related risks; (6) Subjects who are considered not suitable for participating in this clinical trial according to evaluation of investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The global aesthetic improvement scale and facial skin dryness and dull complexion comprehensively improvement | From enrollment to the end of treatment at 3 months

IPD SHARING:
Plan to Share IPD: No